CLINICAL TRIAL: NCT03042247
Title: Prospective Comparison Between FDG-positron Emission Tomography (FDG-PET)/Magnetic Resonance and FDG-PET/Computed Tomography for Staging, Interim Assessment and Restaging in Classical Hodgkin Lymhoma and DLBC Non-Hodgkin Lymphoma
Brief Title: Prospective Comparison Between FDG-PET/MR and FDG-PET/CT in Classical Hodgkin Lymphoma and DLBC Non-Hodgkin Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marco Picardi (Other)
Collaborators: Federico II University (Other)
Responsible Party: Sponsor-Investigator, Marco Picardi, Prof., Federico II University
Organization: Federico II University (Other)
Other Study IDs: FDGMR-LIN
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Diffuse Large B-cell-lymphoma; Classical Hodgkin Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hodgkin lymphoma patients: Hodgkin lymphoma patients with confirmed histological diagnosis
  Interventions: Diagnostic Test: FDG PET/TC and FDG PET/MRI
- DLBC non Hodgkin lymphoma patients: DLBC non Hodgkin lymphoma patients with confirmed histological diagnosis
  Interventions: Diagnostic Test: FDG PET/TC and FDG PET/MRI

INTERVENTIONS:
Diagnostic Test: FDG PET/TC and FDG PET/MRI — Combined assessment with FDG PET/TC and PET/MRI

SUMMARY:
According to the most recent guidelines, total-body imaging techniques are an indispensable element in the staging and post-treatment re-evaluation in patients with lymphoma. Fluorodeoxyglucose-positron emission tomography/computed tomography (FDG-PET/CT) is the gold-standard for the assessment of the disease in these patients. The use of alternative methods, without radiation, such as whole-body magnetic resonance imaging (MRI), could be a valid alternative; this would result an advantage, considering the young age of the majority of patients at diagnosis and the need to undergo to serial assessments. The recent introduction of combined PET total body MRI (PET/MRI) offers the possibility to integrate morphological information with the high resolution of MRI with the metabolic activity of PET, through the uptake of FDG, for a more accurate definition of the extent of disease in patients with lymphoma.

DETAILED DESCRIPTION:
All patients diagnosed with classical Hodgkin lymphoma and diffuse large B-cell non-Hodgkin lymphoma that meet the inclusion criteria will be enrolled in the study. They will undergo an FDG-PET/CT for defining the staging and the therapeutic strategy. PET/MRI scans will be performed immediately upon completion of the PET/contrast-enhanced CT study and FDG tracer will be injected before the PET/CT exam and PET/MRI acquisitions will be practiced using the residual activity of the tracer. All patients will have to provide their informed consent in order to participate in the study.

The combined assessment FDG-PET/CT and FDG-PET/MRI will be performed at diagnosis for staging, at the interim evaluation for early assessment of treatment response after 2 cycles of chemotherapy and finally the post-chemotherapy re-staging. The enrollment period is 24 months for a total of 60 patients with Hodgkin lymphoma and 60 with DLBC non Hodgkin lymphoma.

Patients enrolled in the study will be followed for the diagnostic/therapeutic program at the Hematology Department of Federico II University of Naples, while the FDG-PET/CT and FDG-PET/MRI examinations will be carried out at the IRCSS SDN of Naples. The acquired images will be evaluated by a panel of experienced radiologists and nuclear physicians at the IRCSS SDN Naples.

The results obtained from the examination MRI will not modify in any way the clinical therapeutic choices in the planned chemotherapy for the patient, who will not receive additional radiations. This prospective pilot study will be conducted after approval by the Ethics Committee; each patient will sign an appropriate informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of classical Hodgkin lymphoma and diffuse large B-cell non-Hodgkin lymphoma;
* Age ≥18 years;
* The need of anti-neoplastic treatment;
* Written informed consent;

Exclusion Criteria:

* Carriers of cardiac pacemakers;
* Carriers of metal mesh implants, tissue expanders (breast);
* Holders of metal implants, cochlear implants and stapedial prostheses, plates or screws, wires, nails, spinal-column distractors, ferromagnetic vascular clips, mechanical heart valves, Swan-Ganz catheter, endocorporal electrodes, neurostimulators, vascular filters, stents and metal spirals that they do not know the characteristics (the manufacturer, type and date of implant) and/or secure magnetic compatibility;
* Holders of metal fragments in the eye, visceral or intracranial;
* Tattoo holders executed by less than 6 months;
* Claustrophobic patients;
* Pregnant patients;
* Patients with uncontrolled diabetes mellitus;
* Patients who do not provide written informed consent to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients (>18 yrs) with histological diagnosis of classical Hodgkin lymphoma and non-Hodgkin diffuse large B-cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2021-02-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy in terms of sensitivity and specificity of FDG-PET/MRI in the staging and post-chemotherapy revaluation | 1 year
  Evaluate the diagnostic accuracy in terms of sensitivity and specificity of FDG-PET/MRI in the staging and post-chemotherapy revaluation (early treatment response after 2 cycles of chemotherapy and final assessment) in patients with classical Hodgkin lymphoma and diffuse large B-cell non-Hodgkin lymphoma, as compared to conventional assessment by FDG PET/ contrast-enhanced CT

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Pane, Prof, Principal Investigator — Hematology - AOU Federico II - Naples - Italy; Marco Picardi, Prof, Study Director — Hematology - AOU Federico II - Naples - Italy; Andrea Soricelli, Prof, Study Chair — IRCSS SDN - Naples - Italy
Locations (2):
- Italy (2):
  - Prof Marco Picardi, Naples
  - Prof Marco Picardi - Hematology - AOU FEDERICO II, Napoli

IPD SHARING:
Plan to Share IPD: Undecided